CLINICAL TRIAL: NCT04082338
Title: Long-Term Adherence To Monitoring/Treatment In Underserved Asian Americans With Chronic HBV
Brief Title: Chronic HBV Management for Asian American
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: U54 Liver Cancer Study; 1U54CA221705-01A1 (NIH)
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VPN Toolkit+TM (Experimental): The intervention will be delivered through virtual patient navigation (VPN) toolkit system (a web/mobile application) format.
  Interventions: Behavioral: VPN; Behavioral: TM
- Text Messages (Active Comparator): Receive TM respectively once a week for 5 weeks for every 6 months in the 18-month study period
  Interventions: Behavioral: TM

INTERVENTIONS:
Behavioral: VPN — The intervention will be delivered through virtual patient navigation (VPN) toolkit system (a web/mobile application). The system includes education modules on HBV management, CHB patient success stories and virtual patient navigation clinical support for overcoming barriers.
  In addition to the VPN, each participant will receive 5 text messages; one message once a week for 5 weeks on HBV management for every 6 months in the 18-month study period.
  Arms: VPN Toolkit+TM
Behavioral: TM — Receive TM on HBV management respectively once a week for 5 weeks for every 6 months in the 18-month study period.

SUMMARY:
About 75% of liver cancers are attributed to chronic hepatitis B (CHB). An estimated 2.2 million individuals in the U.S. have CHB. Although Asian Americans make up 6% of total U.S. population, they account for over 58% of Americans with CHB. Prevalence rates of CHB range from 8% to 13% in Asian Americans vs 1% in Non-Hispanic whites (NHW). Asian Americans are 8-13 times more likely to develop liver cancer with 60% higher death rate than NHW. Regular monitoring of CHB is vital in preventing HCC. Research indicates that regular monitoring (e.g., every six months doctor visit; blood tests) combined with antiviral treatment when appropriate, is critical to reduce the risk of liver disease (including HCC). Unfortunately, treatment effectiveness diminishes if CHB patients do not adhere to long-term monitoring and treatment guidelines. Adherence among Asian Americans with CHB is low. Poor healthcare access and significant cultural barriers prevent long-term adherence to monitoring and optimal treatment, placing Asian Americans at disproportionately high risk for HCC and increased healthcare costs.

Building on previous studies, the investigators will use a virtual patient navigation (VPN) toolkit system (a web/mobile application) to help CHB patients improving their liver disease management.

DETAILED DESCRIPTION:
Liver cancer is the second-leading cause of cancer deaths worldwide, which increased at the highest rate of all cancers in the U.S between 2003 and 2012. Asian Americans have the highest incidence and mortality rates of hepatocellular carcinoma (HCC) of all U.S. racial/ethnic groups. About 75% of liver cancers are attributed to chronic hepatitis B (CHB). An estimated 2.2 million individuals in the U.S. have CHB. Although Asian Americans make up 6% of total U.S. population, they account for over 58% of Americans with CHB. Prevalence rates of CHB range from 8% to 13% in Asian Americans vs 1% in Non-Hispanic whites (NHW). Asian Americans are 8-13 times more likely to develop liver cancer with 60% higher death rate than NHW. Regular monitoring of CHB is vital in preventing HCC. Research indicates that regular monitoring (e.g., every six months doctor visit; blood tests) combined with antiviral treatment when appropriate, is critical to reduce the risk of liver disease (including HCC). Unfortunately, treatment effectiveness diminishes if CHB patients do not adhere to long-term monitoring and treatment guidelines. Adherence among Asian Americans with CHB is as low. Poor healthcare access and significant cultural barriers prevent long-term adherence to monitoring and optimal treatment, placing Asian Americans at a disproportionately high risk for HCC and increased healthcare costs.

Building on previous studies, the investigators will use a virtual patient navigation (VPN) toolkit system (a web/mobile application) to help CHB patients improving their liver disease management. This study addresses DHHS and NIH National top priorities, Institute of Medicine's national goal of eliminating HBV and urgent need to evaluate evidence-based interventions that can be integrated into primary care setting and other relevant settings.

The specific aims of the study are:

Aim 1 (Primary) Evaluate comparative effectiveness of Text Message (TM) vs VPN+TM in improving long-term adherence to monitoring (regular doctor visit; blood tests) at 12- and 18- month follow ups. Aim 2 (Secondary) Compare the effectiveness of TM vs VPN+TM in improving and sustaining medication adherence (measured through self-report and electronic monitoring) among Asian Americans with CHB who meet antiviral treatment guidelines. Aim 3 (Exploratory) Examine mediators of intervention effectiveness, including information (knowledge), motivation, and self-efficacy, as well as dose-response.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 and above
* 2. Self-identified Chinese, Korean or Vietnamese ethnicity
* 3. Chronic HBV infection with positive HBV surface antigen (HBsAg)
* 4. Non-compliant to HBV monitoring and treatment guidelines

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grace X Ma, PhD, Principal Investigator — Temple University
Locations (2):
- United States (2):
  - Department of Psychology, Hunter College, New York, New York
  - Center for Asian Health, Lewis Katz School of Medicine, Temple University, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- VPN Toolkit+TM: The intervention will be delivered through virtual patient navigation (VPN) toolkit system (a web/mobile application) format.
  VPN: The intervention will be delivered through virtual patient navigation (VPN) toolkit system (a web/mobile application). The system includes education modules on HBV management, CHB patient success stories and virtual patient navigation clinical support for overcoming barriers.
  In addition to the VPN, each participant will receive 5 text messages; one message once a week for 5 weeks on HBV management for every 6 months in the 18-month study period.
  TM: Receive TM on HBV management respectively once a week for 5 weeks for every 6 months in the 18-month study period.
Period: Overall Study Baseline
Arm/Group | VPN Toolkit+TM | Text Messages
Started | 191 | 191
Completed | 191 | 191
Not Completed | 0 | 0
Period: 12-month Follow-up
Arm/Group | VPN Toolkit+TM | Text Messages
Started | 191 | 191
Completed | 186 | 186
Not Completed | 5 | 5
Period: 18-month Follow-up
Arm/Group | VPN Toolkit+TM | Text Messages
Started | 186 | 186
Completed | 181 | 184
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VPN Toolkit+TM | Text Messages | Total
Number analyzed (Participants) | 191 | 191 | 382
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.29 (0.91) | 53.18 (1.04) | 53.23 (1.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 99 | 198
  Male | 92 | 92 | 184
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Chinese | 148 | 150 | 298
  Vietnamese | 43 | 41 | 84
Born in the US [Count of Participants; unit: Participants]
  Yes | 1 | 4 | 5
  No | 190 | 187 | 377

OUTCOME MEASURES:

1. Primary Outcome: Adherence to Recommended HBV Monitoring: Doctor's Visits
Description: percentage of subjects, who visited doctor's office for HBV at 12-month and 18-month Follow-Up
Time Frame: 12 months, 18 months
Population: There are 3 cases (1 intervention, 2 control cases) missing information on doctor's visit at the 12-month follow-up assessment point.
Measure: Count of Participants; unit: Participants
Arm/Group | VPN Toolkit+TM | Text Messages
Number analyzed (Participants) | 185 | 184
Participants
  Doctor's Visit by 12-month follow-up | 159 | 100
  Doctor's Visit by 18-month follow-up: number analyzed (Participants) | 181 | 184
  Doctor's Visit by 18-month follow-up | 170 | 147

ADVERSE EVENTS:
Time Frame: through study completion, 2 years
Arm/Group | VPN Toolkit+TM | Text Messages
All-Cause Mortality (participants affected / at risk) | 0/191 | 0/191
Serious Adverse Events (participants affected / at risk) | 0/191 | 0/191
Other Adverse Events (participants affected / at risk) | 0/191 | 0/191

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/38/NCT04082338/Prot_SAP_000.pdf